CLINICAL TRIAL: NCT04859387
Title: Effectiveness of Pragmatic Shoulder Techniques in Comparison With Traditional Physical Therapy in Patients With Shoulder Pathologies
Brief Title: Effectiveness of Pragmatic Shoulder Technique VS Traditional Physical Therapy
Acronym: PSTVSTPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helping Hand Institute of Rehabilitation Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rec-2020-F-002
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Pain; Shoulder Impingement; Shoulder Injuries; Frozen Shoulder; Shoulder Capsulitis
Keywords: pragmatic intervention,; shoulder pathologies,; shoulder pain,; shoulder range of motion; pragmatic shoulder intervention,
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Shoulder Injuries; Bursitis

STUDY DESIGN:
Intervention Model Description: quasi-experimental
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): set of pragmatic shoulder techniques
  Interventions: Other: set of pragmatic shoulder technique
- group B (Active Comparator): traditional physical therapy
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Other: set of pragmatic shoulder technique — Group A received pragmatic intervention which includes Pectoralis major and minor stretch, AC joint mobilization, rotator cuff facilitation for subscapularis and infraspinatus, serratus anterior stretch, thoracic manipulation and posterior capsular stretch.
  Arms: group A
Other: traditional physical therapy — Group B received traditional interventions which includes modalities such as TENS and hot pack, soft tissue mobilization, joint mobilization, stretching and strengthening etc. other than pragmatic intervention
  Arms: group B

SUMMARY:
Isolated and combined effectiveness of pragmatic protocols on shoulder range of motion had been investigated and found effective in healthy participants. To our knowledge, there was insufficient literature to support the comparison between pragmatic and traditional protocols in the treatment of shoulder pathologies.

DETAILED DESCRIPTION:
Different physical therapy treatments are being used for shoulder pathologies which include modalities (hot pack, TENS), ROM exercises, stretching, strengthening, soft tissue mobilization and set of pragmatic manual techniques.The set of pragmatic manual therapies are novel techniques (comprises of acromioclavicular mobilization, serratus anterior stretch, thoracic manipulation, RC facilitation, and PCS) and its isolated effectiveness on ROM in healthy subjects has been investigated and found effective. These studies recommended the use of a pragmatic protocol for the prevention and rehabilitation of shoulder injuries and pathologies (unpublished data).As per our knowledge there is insufficient literature to support the comparison of the effectiveness of a set of pragmatic protocols with traditional interventions. Our research is proposed to compare the efficacy of pragmatic interventions with that of traditional interventions in patients with shoulder pathology and their effect on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Functional movement score 1 and 2 or limitation in Range of motion of Abduction, internal rotation, external rotation, RUBB, and RDBN. All or only one of the limitations in comparison with the unaffected shoulder joint.

Exclusion Criteria:

* Patients with shoulder instability. Functional movement score 3 and 0. Individuals with recent fractures of fewer than 6 weeks duration. Cancerous Growth around the shoulder girdle. Breast cancer and undergoing chemotherapy and radiotherapy. RA arthritis patients. Long-term use of steroids and severe osteoporosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
shoulder Range of motion | 5 days
  will be measured in degrees by digital inclinometer
functional movements | 5 days
  will be measured in centimeters by inchi tape

CONTACTS AND LOCATIONS:
Overall Officials: Keramat Ullah Keramat, Ph.D*, Principal Investigator — HHIRS Trust
Locations (1):
- Helping hand Institute of Rehabilitation Sciences Trust, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
as per the decision of helping hand research ethical committee (HHREC)

REFERENCES:
- [Background] Keramat KU, Naveed Babur M. Pragmatic posterior capsular stretch and its effects on shoulder joint range of motion. BMJ Open Sport Exerc Med. 2020 Sep 9;6(1):e000805. doi: 10.1136/bmjsem-2020-000805. eCollection 2020. PMID 33062302
- [Background] Keramat KU, Babar MN. Serratus Anterior Stretch: A Novel Intervention and Its Effect on the Shoulder Range of Motion. J Sport Rehabil. 2021 Jan 8;30(5):824-827. doi: 10.1123/jsr.2020-0121. PMID 33418538